CLINICAL TRIAL: NCT00020865
Title: Multicenter, Double-Blind, Randomized Study to Compare the Safety and Efficacy of Levofloxacin With That of Cefepime in the Treatment of Fever and Neutropenia - Phase IIIB
Brief Title: Levofloxacin Compared With Cefepime in Treating Cancer Patients With Fever and Neutropenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000068726; UCLA-0006093; MCNEIL-CAPSS-118; NCI-G01-1965
Record Dates: First submitted 2001-07-11; First posted 2004-03-17 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-05

CONDITIONS: Fever, Sweats, and Hot Flashes; Infection; Leukemia; Lymphoma; Neutropenia; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; fever, sweats, and hot flashes; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; primary central nervous system non-Hodgkin lymphoma; neutropenia; infection; prolymphocytic leukemia; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; intraocular lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Fever; Hot Flashes; Infections; Leukemia; Lymphoma; Neutropenia; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Hairy Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone | interventions — Cefepime; Levofloxacin

INTERVENTIONS:
Drug: cefepime hydrochloride
Drug: levofloxacin

SUMMARY:
RATIONALE: Levofloxacin may be effective in reducing fever and controlling other symptoms of neutropenia in patients who are being treated for cancer. It is not yet known whether levofloxacin is more effective than cefepime in reducing fever and controlling symptoms of neutropenia.

PURPOSE: Randomized phase III trial to compare the effectiveness of levofloxacin with that of cefepime in reducing fever and controlling symptoms of neutropenia in patients who are being treated for cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the safety and efficacy of levofloxacin versus cefepime in cancer patients with fever and neutropenia. II. Compare the percentage of patients whose fever defervesces and who have no signs or symptoms of infection with and without therapeutic modification. III. Compare the percentage of survival of patients treated with these 2 regimens with no therapeutic modifications. IV. Compare the overall survival of patients treated with these 2 regimens regardless of therapeutic modifications. V. Compare the time to resolution of fever in patients treated with these regimens. VI. Compare the microbiologic response by pathogen and site of infection in patients treated with these regimens. VII. Compare the percentage of patients whose fever defervesces only after resolution of neutropenia (absolute neutrophil count at least 500/mm3) with no therapeutic modification.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to type of malignancy (solid tumor, including lymphoma vs leukemia), prior prophylactic antibiotics (yes vs no), and participating center. Patients are randomized to one of two treatment arms. Arm I: Patients receive levofloxacin IV over 90 minutes once daily for 14-28 days. Arm II: Patients receive cefepime IV over 30 minutes every 8 hours for 14-28 days. Patients may receive additional antifungal, antibacterial, or antiviral therapy if condition has deteriorated, no response is seen in 72 hours, or and infection is suspected or documented. Patients are followed at 1-3 and 7-12 days and then at 3-4 weeks.

PROJECTED ACCRUAL: Approximately 260-400 patients (130-200 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of malignancy Solid tumor (including lymphoma) or leukemia Hospitalized and anticipated to remain hospitalized during study Febrile defined as oral temperature of at least 100.4 degrees F (38 degrees C) on 2 occasions within 24 hours OR at least 100.8 degrees F (38.2 degrees C) on a single reading No obvious noninfectious cause of fever (e.g., platelet transfusion) Neutropenic, defined as absolute neutrophil count (ANC) currently less than 500/mm3 OR anticipated to be less than 500/mm3 within 24 hours of study entry Anticipated ANC to be less than 500/mm3 for at least 72 hours No neutropenia unassociated with malignancy No chronic neutropenia No neutropenia anticipated to last more than 14 days No acute myelogenous leukemia unless receiving consolidation chemotherapy or induction dose that does not prolong neutropenia for more than 3 weeks No infection due to an identified organism No high likelihood of infection due to anaerobic organisms, including intra-abdominal infections or perirectal abscess at admission No known osteomyelitis No requirement for new antifungal agent

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: At least 14 days Hematopoietic: See Disease Characteristics Hepatic: Not specified Renal: Creatinine clearance at least 20 mL/min No oliguria (urine output less than 20 mL/hour) unresponsive to fluid challenge Cardiovascular: No shock or hypotension (supine systolic blood pressure less than 80 mmHg) unresponsive to fluid challenge Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No HIV infection with CD4 counts less than 200/mm3 No significant risk for seizures No unstable psychiatric disorder Weight greater than 40 kg No prior allergic or severe adverse reaction to study drugs or to any member of the quinolone or beta-lactam class of antibacterials No disorder or disease that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior sargramostim (GM-CSF) or filgrastim (G-CSF) for current course of chemotherapy Concurrent GM-CSF or G-CSF allowed if neutropenia lasts at least 3 days Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No prior treatment under this protocol No prior prophylactic anti-infectives other than acyclovir or sulfamethoxazole with trimethoprim At least 72 hours since prior systemic antibiotics (except prophylactic sulfamethoxazole with trimethoprim) At least 30 days since prior experimental drug or medical device (except drugs currently marketed in the United States for the treatment of the malignancy) No other concurrent systemic antibacterial agents No concurrent topical antimicrobial agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09

CONTACTS AND LOCATIONS:
Overall Officials: Mary C. Territo, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States